CLINICAL TRIAL: NCT03744416
Title: Effectiveness of a Counseling Intervention in the Birth Plan for Pregnant Women (APLANT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Catalan Institute of Health (Other Government); University of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4R17/085-1
Record Dates: First submitted 2018-10-23; First posted 2018-11-16 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2019-08

CONDITIONS: Birth; Satisfaction
Keywords: birth plan; share decision making; pregnant women; midwife; satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Cluster randomised trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Counseling based on Epstein's active decision making on birth plan
  Interventions: Other: Counseling based on Epstein's active decision making
- Control group (No Intervention): The standard midwife's advice on birth plan during prenatal care.

INTERVENTIONS:
Other: Counseling based on Epstein's active decision making — Birth information leaflet. Based on the best evidence practice. Midwives' training on share decision making based on Epstein model. Pregnant intervention. The pregnant women will receive from the midwives the birth plan (BP) in the prenatal check at the health center, between the 24-28 weeks, to be completed at home. Later, on the visit between 29-33 weeks, the midwives will provide the "birth information leaflet" and carry out the counseling intervention based on "shared decision making" to the pregnant women. As well, midwives will deliver a second BP that pregnant woman will fill at home. On the prenatal check between 34 to 40 weeks, the midwife will save a copy of the latest BP. The midwife will instruct the woman to deliver the BP when she arrives to the hospital for birth.
  Arms: Intervention group

SUMMARY:
This study assesses the effectiveness of a birt plan (BP) counseling intervention in pregnant women.

Half of the pregnant women receive the intervention and the other half receive the usual practice

DETAILED DESCRIPTION:
The birth plan (BP) is the written expression of the preferences of the pregnant woman about the management of her birth, in those cares in which there are equally effective and safe alternatives. In Spain, it was introduced into the National Health System when the "Normal Birth Attention Strategy" was developed, and in Catalonia when the Department of Health published the "Protocol to the natural assistance of normal childbirth", all with the purpose of responding to the demand of women to participate actively in their birth. Its main purpose is to promote decision-making not influenced by the emotions that arise during the birth process and to provide a communication vehicle between the future parents, the care provider and the hospital team. In addition, it allows pregnant women to understand their personal values, needs and concerns in the process of birth. The preparation of the BP can help the pregnant woman to have real expectations of childbirth, make her involved in the decision making process, thus increasing control over the birth process and having a satisfactory experience with the experience of childbirth .

Studies on the impact of the birth plan in reference on the satisfaction of women in childbirth, on obstetric outcomes and on the perception that women and professionals have of them, are scarce and inconclusive. Observational studies related that the use of BP was associated with an increase in: normal birth, late clamping of the umbilical cord, the realization of skin with skin and less use of epidural analgesia. In addition, there are researches with quantitative and qualitative methodology in which they relate the fulfillment of the BP with a greater satisfaction of the women, a greater fulfillment of the expectations and a better control of the delivery. However, others studies they do not relate it to a higher delivery satisfaction. There is also disparity between the views of midwives and women on the utility of the effect of BP on obstetric outcomes In 2016 a survey carried out in Catalonia on the satisfaction of women in the care of the maternity process showed that the overall level of satisfaction with the care received was high, 8.30 out of 10. However, women only refer who received sufficient information in pregnancy, delivery and postpartum in 67.2%, 64.2% and 57.6% respectively.

Of the different models of care relationship, the deliberative model focuses on joint collaborative work between patient and professional, in which the dialogue has a central role and shared decision-making (SDM) is present in said model . There is a large bibliography on the definition of SDM, as well as the elements that should be present in this process. According to Epstein et al, clinical decision making should be approached from the creation of a collaborative relationship with the patient and family using the best available evidence, consistent with the values, objectives and capacities of the patients. The use of decision support tools, such as support material, can help health professionals to provide information and advice on options during pregnancy and to support women in shared decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with prenatal in the study centers
* Birth in the reference hospitals.

Exclusion Criteria:

* Illiteracy
* Language barrier
* Very high risk pregnancy
* Drug addiction
* Alcoholism,
* Heart disease: grade 2, 3 and 4,
* Serious associated maternal pathology,
* Type I-II diabetes,
* Uterine malformation,
* Diagnosed fetal malformation,
* Threat of premature birth,
* Twin or multiple gestation,
* Cervical incompetence,
* previous history perinatal death,
* Intrauterine growth retardation,
* Previous placenta,
* Isoimmunization,
* Mild-severe preeclampsia,
* several maternal infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Delivery of the birth plan in hospital | 6 weeks postpartum
  Nominal scale: yes, no
Sufficient information received in pregnancy about childbirth. | 6 weeks postpartum
  Nominal scale: yes, no
Overall satisfaction at birth and satisfaction in the degree of participation in the decision making in the first and second stage of labor. | 6 weeks postpartum
  Satisfaction Childbirth Rating Scale validate. Likert scale: very dissatisfied; little satisfied; indifferent; satisfied; very satisfied.

SECONDARY OUTCOMES:
Reasons for non-delivery the birth plan in the hospital: | 6 weeks postpartum
  Nominal scale: I thought it was not necessary, I forgot, the professionals who attended me did not ask me, others.
Preferences for childbirth care expressed in birth plan. | Until birth
  Birth plan questionnaires. Descriptive scale. Preferences related to: procedures, pain relief methods, care during the first and second stage period, newborn care and breastfeeding
Degree of usefulness of the completion of the birth plan | 6 weeks postpartum
  Scale likert from 0 to 5 : 0 is nothing useful, little useful, indifferent, quite useful 5 very useful.
Use of the birth plan in the following pregnancy | 6 weeks postpartum
  Nominal scale: Yes, no.

CONTACTS AND LOCATIONS:
Overall Officials: Encarnación López-Gimeno, Principal Investigator — Catalan Institute of Health; Gemma Falguera-Puig, PhD, Study Director — Catalan Institute of Health; Gloria Seguranyes, PhD, Study Director — University of Barcelona
Locations (4):
- Spain (4):
  - Catalan Health Institute, Badalona, Barcelona
  - Catalan Health Institute, Granollers, Barcelona
  - Catalan Health Institute, Mollet del Vallès, Barcelona
  - Catalan Health Institute, Barcelona

IPD SHARING:
Plan to Share IPD: No